CLINICAL TRIAL: NCT03479294
Title: Real-World Study on Adjuvant Therapy Combined With Shenlingcao Oral Liquid in Patients for Stage II and IIIA Non-small Cell Lung Cancer After Radical Resection
Status: Terminated | Type: Observational
Why Stopped: Because of the difficulty of research operation, we changed to another research design.
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Sun Xin, Director, West China Hospital
Other Study IDs: 320.6750.17576
Record Dates: First submitted 2018-03-19; First posted 2018-03-27 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Chemotherapy, Adjuvant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: Exposure group patients are those who voluntarily choose to use Shenlingcao Oral Liquid recommended by the doctor in NSCLC patients receiving adjuvant chemotherapy. Jiangzhong Group will donate the first 30 bottles of medicine, and afterwards, patients may purchase if they still need to take it. The length of time and dose of Shenlingcao Oral Liquid are unlimited and other adjunctive treatments may be used at the same time.
  Interventions: Drug: Shenlingcao Oral Liquid
- Control group: Control group patients are those who voluntarily choose not to use Shenlingcao Oral Liquid recommended by the doctor in NSCLC patients receiving adjuvant chemotherapy.

INTERVENTIONS:
Drug: Shenlingcao Oral Liquid — Shenlingcao Oral Liquid is a health product, and its main components are American ginseng, lucidum, Cordyceps fermented powder Cs-4, rose, maltitol and water. Shenlingcao Oral Liquid can relieve physical fatigue and enhance immunity.
  Groups: Exposure group

SUMMARY:
This study will establish a multi-center, prospective registration database. The included population are stage II and IIIA NSCLC patients undergoing R0 resection and will be scheduled for adjuvant chemotherapy. Before the first adjuvant chemotherapy, under the recommendation of a doctor, patients will voluntarily choose to use (exposed group) or not to use (control group) Shenlingcao Oral Liquid, which donated by Jiangzhong Group for 30 bottles. The research centers need to be consecutively enrolled patients according to the allocation of the number of cases according to the ratio of 3: 1 in exposure group and control group.

The exposed and control groups will be followed up to 36 months (non-allelic follow-up). Information from patients will be prospectively collected, including baseline, chemoradiation, use of Shenlingcao Oral Liquid and the other complementary drugs, and various outcome measures (the questionnaire of EORTC QLQ, death, tumor recurrence, tumor metastasis, and chemotherapy-induced side effects of the blood system, etc.). Follow-up points included: Baseline (before giving chemotherapy), 2-3 days after each chemotherapy cycle, and 6,12,18,24,30,36 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older;
* Pathological diagnosis of patients with stage II, III A primary NSCLC;
* R0 resection has been accepted;
* Received adjuvant chemotherapy or adjuvant chemotherapy for the first time after surgery;
* Informed consent has been signed.

Exclusion Criteria:

* Incorporation of other malignant tumors (such as leukemia, liver cancer, etc.)；
* Patients with unclear pathological types；
* Patients with unclear pathological staging；
* Preserved Shenlingcao Oral Liquid before R0 resection surgery；
* Received immunotherapy or targeted therapy before R0 resection surgery；
* Radiotherapy and chemotherapy before R0 resection surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing adjuvant radiotherapy or chemotherapy for Stage II and IIIA Non-small Cell Lung Cancer After Radical Resection
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
The quality of life | About 20 minutes
  A scale for the quality of life of cancer patients developed by the European Organization for Research and Treatment (according to EORTC QLQ-C30 V3.0)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, Principal Investigator — The Chinese Cochrane Center，West China Hospital, Sichuan University
Locations (1):
- Tianjin Chest Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided